CLINICAL TRIAL: NCT00281840
Title: A Phase II Study of Bevacizumab in Combination With Docetaxel and Radiation in Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Bevacizumab, Docetaxel, and Radiation Therapy in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6304; P30CA043703 (NIH); CASE6304 (Other: Case Comprehensive Cancer Center); 03-05-50 (Other: University Hospitals IRB)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Bevacizumab; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab with docetaxel and radiation therapy (Experimental)
  Interventions: Biological: bevacizumab; Drug: docetaxel; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab — Bevacizumab IV over 30-90 minutes once every 2 weeks for up to 1 year. Bevacizumab, which stops 8 weeks before surgery, may restart 4 weeks after surgery and continue for 9 months in the absence of disease progression or unacceptable toxicity.
Drug: docetaxel — docetaxel IV over 1 hour once a week for 8 weeks
Procedure: conventional surgery — 8-10 weeks after the completion of chemoradiotherapy, patients may undergo neck dissection
Radiation: radiation therapy — radiotherapy once daily, 5 days a week, for 8 weeks

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bevacizumab together with docetaxel and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with docetaxel and radiation therapy works in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in patients with stage III or IV squamous cell carcinoma of the head and neck treated with bevacizumab in combination with docetaxel and radiotherapy.

Secondary

* Compare the objective response rate, locoregional control rate, duration of response, patterns of failure, and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients undergo radiotherapy once daily, 5 days a week, for 8 weeks and receive docetaxel IV over 1 hour once a week for 8 weeks. Patients also receive bevacizumab IV over 30-90 minutes once every 2 weeks for up to 1 year.

Approximately 8-10 weeks after the completion of chemoradiotherapy, patients may undergo neck dissection. Bevacizumab, which stops 8 weeks before surgery, may restart 4 weeks after surgery and continue for 9 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck

  * Stage III or IV disease

    * No evidence of distant metastases
  * No salivary gland or paranasal sinus squamous cell carcinoma
* No disease with close proximity to a major vessel
* Measurable disease
* No known CNS or brain metastases

  * Patients with intracranial extension without cerebral involvement may be eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* AST and ALT ≤ 2 times upper limit of normal
* PT normal
* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min
* Urine protein: creatinine ratio < 1.0
* No bleeding diathesis or coagulopathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No pre-existing peripheral neuropathy ≥ grade 2
* No ongoing or active infection
* No serious non-healing wound, ulcer, or bone fracture
* No New York Heart Association class II-IV congestive heart failure
* No significant arrhythmias requiring medication
* No myocardial infarction within the past 6 months
* No stroke within the past 6 months
* No symptomatic coronary artery disease
* No second- or third-degree heart block or bundle branch block
* No unstable angina pectoris
* No hypertension (i.e., blood pressure ≥ 150/100 mm Hg)
* No other clinically significant heart disease
* No significant traumatic injury within the past 4 weeks
* No psychiatric illness or social situation that would preclude study compliance
* No HIV positivity
* No other malignancy within the past 5 years except squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No other uncontrolled illness
* No poorly compliant patients

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No prior investigational anticancer agents
* More than 4 weeks since prior major surgery
* More than 1 week since prior minor surgery, fine-needle aspiration, or core needle biopsy
* No concurrent major surgery except planned neck dissection
* No concurrent routine colony-stimulating factor therapy
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Savvides, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (6):
- United States (6):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - UHHS Chagrin Highlands Medical Center, Orange Villager, Ohio
  - UHHS Westlake Medical Center, Westlaker, Ohio
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Yao M, Galanopoulos N, Lavertu P, Fu P, Gibson M, Argiris A, Rezaee R, Zender C, Wasman J, Machtay M, Savvides P. Phase II study of bevacizumab in combination with docetaxel and radiation in locally advanced squamous cell carcinoma of the head and neck. Head Neck. 2015 Nov;37(11):1665-71. doi: 10.1002/hed.23813. Epub 2014 Oct 29. PMID 24954745
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=case6304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from University Hospitals (Cleveland OH) and University of Pittsburgh (Pittsburgh PA) from September 2005 through September 2008.
Groups:
- Bevacizumab With Docetaxel and Radiation Therapy: Radiation therapy will be delivered using standard once-daily fractionation, five days a week for 8 weeks. Bevacizumab is administered intravenously once on day 1 every two weeks during the course of radiation and up to one year following completion of radiation therapy, at which point bevacizumab will be discontinued.Patients meeting planned neck dissection criteria, will not receive bevacizumab therapy following completion of concurrent chemo-radiation therapy (for at least 8 weeks prior to surgery). Bevacizumab therapy will restart 4 weeks after planned neck dissection for nine months.Docetaxel is administered intravenously once per week only during the course of radiation.
Period: Overall Study
Arm/Group | Bevacizumab With Docetaxel and Radiation Therapy
Started | 30
Completed | 5
Not Completed | 25
Not completed — Adverse Event | 12
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 3
Not completed — Disease Progression | 2
Not completed — exceed maximum delay in treatment | 1
Not completed — Complicating Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab With Docetaxel and Radiation Therapy
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  40-49 years | 4
  50-59 years | 16
  60-69 years | 9
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: The time to disease progression is calculated from the date of treatment. Data for patients who remain disease progression free are censored as of date when the last follow-up information is obtained.
Time Frame: 5 yrs after treatment
Population: Patients who received at least one treatment on study
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab With Docetaxel and Radiation Therapy
Number analyzed (Participants) | 30
Months | 44.2 [33.79 to 54.61]

2. Secondary Outcome: Response Rate
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence. The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST). A response will be determined by at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
Time Frame: 5 years
Population: Patients with evaluable tumors at the end of the study
Measure: Number; unit: participants
Arm/Group | Bevacizumab With Docetaxel and Radiation Therapy
Number analyzed (Participants) | 26
participants
  Complete Response | 16
  Partial Response | 6
  Progressive Disease | 1
  Stable Disease | 3

ADVERSE EVENTS:
Arm/Group | Bevacizumab With Docetaxel and Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab With Docetaxel and Radiation Therapy (N=30)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Wound-Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (3)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 3 (3)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 1 (1) — map to v4.0 as vascular disorder (other)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — not due to neuropathy
Abdominal pain or cramping (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine (Renal and urinary disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab With Docetaxel and Radiation Therapy (N=30)
Constipation (Gastrointestinal disorders) | 20 (39)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 20 (46)
Mouth dryness (Gastrointestinal disorders) | 19 (28)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 19 (41)
Nausea (Gastrointestinal disorders) | 18 (33)
Anorexia (Gastrointestinal disorders) | 15 (31)
Mucositis due to radiation (Gastrointestinal disorders) | 15 (31)
Vomiting (Gastrointestinal disorders) | 14 (22)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 12 (19)
Gastrointestinal (congestion) (Gastrointestinal disorders) | 9 (12)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 9 (18)
Salivary gland changes (Gastrointestinal disorders) | 8 (13)
Dehydration (Gastrointestinal disorders) | 6 (13)
Dysphagia-pharyngeal related to radiation (Gastrointestinal disorders) | 5 (11)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 29 (54)
Weight loss (General disorders) | 29 (61)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 9 (10)
Rigors, chills (General disorders) | 6 (6)
Sweating (diaphoresis) (General disorders) | 4 (4)
Constitutional Symptoms (General disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 27 (58)
Hyperglycemia (Metabolism and nutrition disorders) | 26 (96)
Hypocalcemia (Metabolism and nutrition disorders) | 17 (45)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (13)
Hypokalemia (Metabolism and nutrition disorders) | 8 (27)
Hypermagnesemia (Metabolism and nutrition disorders) | 7 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hemoglobin (Blood and lymphatic system disorders) | 26 (55)
Lymphopenia (Blood and lymphatic system disorders) | 26 (158)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7 (13)
Platelets (Blood and lymphatic system disorders) | 3 (3)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 23 (40)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (9)
Dermatology/Skin (erythema) (Skin and subcutaneous tissue disorders) | 4 (4) — Erythema at PEG, neck erythema, abrasions from fall, neck fibrosis
Flushing (Skin and subcutaneous tissue disorders) | 4 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 22 (55)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 15 (26)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 13 (25)
Alkaline phosphatase (Investigations) | 7 (11)
Bilirubin (Investigations) | 4 (8)
Pain (General disorders) | 26 (71)
Headache (Nervous system disorders) | 4 (4)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 3 (4)
Chest pain (non-cardiac and non-pleuritic) (Cardiac disorders) | 3 (3)
Earache (otalgia) (Ear and labyrinth disorders) | 3 (4)
Pain due to radiation (Injury, poisoning and procedural complications) | 3 (3)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (3)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 17 (27)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 10 (12)
Neuropathy-sensory (Nervous system disorders) | 10 (14)
Mood alteration-depression (Psychiatric disorders) | 9 (10)
Dizziness/lightheadedness (Nervous system disorders) | 6 (6)
Confusion (Psychiatric disorders) | 4 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infection without neutropenia (Infections and infestations) | 12 (22)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (10)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 3 (5)
Creatinine (Investigations) | 4 (11)
Proteinuria (Renal and urinary disorders) | 4 (7)
Incontinence (Renal and urinary disorders) | 2 (3)
Edema (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 7 (7)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Hemorrhage (bloody nose) (Vascular disorders) | 2 (2)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 2 (3)
Hot flashes/flushes (Vascular disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3)
Auditory/Hearing (hard of hearing) (Ear and labyrinth disorders) | 4 (4)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (3)
Partial thromboplastin time (PTT) (Investigations) | 2 (2)
Prothrombin time (PT) (Investigations) | 2 (2)
Vision-blurred vision (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes